CLINICAL TRIAL: NCT05638464
Title: Multisite Transcranial Direct Current Stimulation Targeting Motor Network by Mapping Electric Fields With Task-based fMRI to Promote Hand Function Recovery After Stroke
Brief Title: Multisite Transcranial Direct Current Stimulation to Promote Hand Function Recovery After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor and Chairman, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018.661
Record Dates: First submitted 2022-11-16; First posted 2022-12-06 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multisite HD-tDCS with EMG-driven robot hand group (Experimental): The stimulation electrodes are fixed on the ipsilesional sensorimotor cortex according to the brain activation map detected by task based fMRI.
  Interventions: Device: multisite HD-tDCS EMG-driven robot hand
- Sham HD-tDCS EMG-driven robot hand group (Sham Comparator): The stimulator will be applied for 20 minutes with only 30s ramp-up and ramp-down stimulation delivered.
  Interventions: Device: Sham HD-tDCS EMG-driven robot hand

INTERVENTIONS:
Device: multisite HD-tDCS EMG-driven robot hand — Multisite HD-tDCS will individual stimulation montages with robot hand training will be applied on chronic stroke survivors. In the multisite HD-tDCS group, 5-8 sintered Ag/AgCl ring electrodes will be placed based on the neuroimaging and computation modelling. The location of the electrodes will be identified by the individual brain activity in the primary motor cortex derived from tasked-based fMRI. The Finite Element Model (FEM) will be used to simulate the electric field distribution on individual brain. Optimization of stimulation montages will be based on the derived activation pattern of the brain. After 20-minute multisite HD-tDCS, EMG-driven robot hand training will be conducted.
  Arms: multisite HD-tDCS with EMG-driven robot hand group
Device: Sham HD-tDCS EMG-driven robot hand — Sham stimulation with robot hand training will be applied on chronic stroke survivors.
  After the sham stimulation, EMG-driven robot hand training will be conducted.
  Arms: Sham HD-tDCS EMG-driven robot hand group

SUMMARY:
A novel multisite high definition tDCS (HD-tDCS) in healthy people showed that such network-targeted stimulation could enhance motor excitability beyond traditional stimulation which targeting only one region. It showed that the excitability following multisite HD-tDCS was more than double the increase following conventional tDCS. To consider the various lesion site of different stroke survivors. The electrode placements based on personalized lesion profiles and anatomical features can be determined using finite element modeling, with lesion profiles generated from fMRI and advanced algorithms calculating the current density to maximize the modulation effect. Combining motor network interaction and the new multisite electrode montage may further provide a potential to facilitate stroke recovery.

ELIGIBILITY:
Inclusion Criteria:

* first-ever stroke, the duration after stroke exceeds 12 months;
* mild to moderate upper extremity motor function deficit, determined by the Fugl-meyer assessment of upper extremity (FMAUE) scores between 15 and 53;
* detectable voluntary muscle sEMG signal from flexor digitorum (FD) and extensor digitorum (ED);
* scored below 3 in the Modified Ashworh Score (MAS) of FD and ED;
* sufficient cognitive function to follow the assessment and training instructions, determined by Mini Mental State Examination score of more than 21.

Exclusion Criteria:

* history of epilepsy, or any other contradictions of brain stimulation;
* severe joint contracture of elbow or shoulder, or pain induced by any other neurological, neuromuscular, and orthopedic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity | 6-month after intervention
  It is used to evaluate and measure upper-limb recovery in post-stroke hemiplegic patients, and items are scored on a 3-point ordinal scale

SECONDARY OUTCOMES:
Action Research Arm Test | 6-month after intervention
  The ARAT is a 19-item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement) to assess upper limb functioning
Magnetic Resonance Imaging (MRI) | 6-month after intervention
  It is used to identify neural correlates of stimulation-induced behavioral gains for investigating tDCS-induced changes in brain activations
Electroencephalography (EEG) | 6-month after intervention
  It is used to investigate the changes in corticomuscular coherence for studying connectivity between the brainwave using EEG and the affected hand muscles using EMG.
Electromyography (EMG) | 6-month after intervention
  EMG will be used to detect muscle activation change and muscle co-contraction pattern alteration.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kai-yu Tong, PhD, Principal Investigator — Department of Biomedical Engineering, CUHK
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Hu C, Ti CHE, Yuan K, Chen C, Khan A, Shi X, Chu WC, Tong RK. Effects of high-definition tDCS targeting individual motor hotspot with EMG-driven robotic hand training on upper extremity motor function: a pilot randomized controlled trial. J Neuroeng Rehabil. 2024 Sep 20;21(1):169. doi: 10.1186/s12984-024-01468-w. PMID 39304930